CLINICAL TRIAL: NCT00958438
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of Rilonacept for the Prophylaxis of Gout Flares During the Initiation of Allopurinol Therapy
Brief Title: PREventative Study Against URate-Lowering Drug-Induced Gout Exacerbations (PRE-SURGE 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-GA-0816; 2008-007762-39 (EudraCT Number)
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Gout
Keywords: Intercritical Gout; Metabolism, Inborn Errors; Allopurinol; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Metabolic disorder; Purine-Pyrimidine Metabolism, Inborn Errors; Gout
MeSH Terms: conditions — Gout; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases; Purine-Pyrimidine Metabolism, Inborn Errors | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Two subcutaneous injections of Placebo (for Rilonacept ) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 15.
  Interventions: Drug: Placebo
- Rilonacept 80 mg (Experimental): Two subcutaneous injections of Rilonacept 80 mg (for a total of 160 mg) as a loading dose on Day 1, followed by a single 80 mg injection of Rilonacept qw from Week 1 to Week 15.
  Interventions: Drug: Rilonacept
- Rilonacept 160 mg (Experimental): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) as a loading dose on Day 1, followed by a single 160 mg injection of Rilonacept qw from Week 1 to Week 15.
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Placebo — Placebo loading dose followed by placebo subcutaneous (SC) injection (2 mL) once a week for 16 weeks.
  Arms: Placebo
Drug: Rilonacept — Rilonacept 160 mg SC loading dose followed by Rilonacept 80 mg/2 mL SC injections once a week for 16 weeks.
  Arms: Rilonacept 80 mg
Drug: Rilonacept — Rilonacept 320 mg SC loading dose followed by Rilonacept 160 mg/2 mL SC injections once a week for 16 weeks.
  Arms: Rilonacept 160 mg

SUMMARY:
The purpose of this clinical research study was to determine the safety and effectiveness of an experimental drug called rilonacept in participants with gout who are beginning allopurinol treatment for gout. Participants will participate in this study for approximately 22 weeks. Rilonacept was being studied for use in preventing allopurinol-induced gout flares.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 80 years of age;
* Previously met the preliminary criteria of the American Rheumatism Association (ARA) for the classification of the acute arthritis of primary gout;
* At least 2 gout flares in the year prior to the screening visit;
* Serum uric acid greater than or equal to 7.5 mg/dL at the screening visit.

Exclusion Criteria:

* Acute gout flare within 2 weeks of the screening visit or during screening;
* Persistent chronic or active infections;
* History of an allergic reaction to allopurinol;
* History or presence of cancer within 5 years of the screening visit;
* Previous exposure to Rilonacept;
* Use of allopurinol, benzbromarone, febuxostat, probenecid or sulfinpyrazone within 3 months prior to the screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Evans, PharmD, Study Director — Regeneron Pharmaceuticals
Locations (61):
- Germany (11):
  - Berlin
  - Essen
  - Goch
  - Hamburg
  - Kassel
  - Künzing
  - Lollar
  - Magdeburg
  - München
  - Rhaunen
  - Siegen
- India (10):
  - Ahmedabad
  - Bangalore
  - Gandhinagar
  - Hyderabaad
  - Kolkata
  - Mangalore
  - Pune
  - Secunderabad
  - Vadodara
  - Varanasi
- Indonesia (8):
  - Denpasar
  - Jakarta
  - Kemerdekaan
  - Palembang
  - Semarang
  - South Sulawesi
  - West Java
  - Yogyakarta
- South Africa (23):
  - Benoni
  - Bloemfontein
  - Breyten
  - Cape Town
  - Dundee
  - Durban
  - Durban North
  - eManzimtoti
  - Gauteng
  - Johannesburg
  - Kempton Park
  - Krugersdorp
  - KZ-Natal
  - Lenasia
  - Lyttleton
  - Middleburg
  - Port Elizabeth
  - Pretoria
  - Roodepoort
  - Scottburgh
  - Somerset West
  - Soweto
  - Worcester
- Taiwan (9):
  - Yungkang City, Tainan
  - Changhua
  - Dalin Town
  - Hualien City
  - Kaohsiung City
  - Kwei-Shan
  - Taichung
  - Tainan
  - Taipei

REFERENCES:
- [Derived] Mitha E, Schumacher HR, Fouche L, Luo SF, Weinstein SP, Yancopoulos GD, Wang J, King-Davis S, Evans RR. Rilonacept for gout flare prevention during initiation of uric acid-lowering therapy: results from the PRESURGE-2 international, phase 3, randomized, placebo-controlled trial. Rheumatology (Oxford). 2013 Jul;52(7):1285-92. doi: 10.1093/rheumatology/ket114. Epub 2013 Mar 13. PMID 23485476
- See also: Rilonacept — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=501081761&QV1=RILONACEPT
- See also: Allopurinol — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=000315300&QV1=ALLOPURINOL
- See also: Allopurinol sodium — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=017795210&QV1=ALLOPURINOL+SODIUM

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 57 study sites in European Union (EU) and rest of world (ROW) between 7 March 2009 and 17 December 2010. A total of 471 participants were screened in the study.
Pre-assignment Details: Out of 471 participants, 248 were randomized and treated in the study. Participants were randomized in 1:1:1 ratio to receive Placebo or Rilonacept 80 mg or Rilonacept 160 mg.
Period: Overall Study
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Started | 82 | 82 | 84
Completed | 72 | 72 | 78
Not Completed | 10 | 10 | 6
Not completed — Protocol Violation | 3 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 1
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Other than specified above | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg | Total
Number analyzed (Participants) | 82 | 82 | 84 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.87) | 52.6 (11.47) | 49 (11.77) | 51.1 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 17
  Male | 77 | 77 | 77 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 82 | 82 | 84 | 248
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 29 | 23 | 30 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 14 | 10 | 34
  White | 43 | 45 | 44 | 132
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Gout Flares Per Participant Assessed From Day 1 to Day 113 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flares per participant was reported for this outcome measure.
Time Frame: Day 1 to Day 113 (Week 16)
Population: Full analysis set (FAS) that included all randomized participants who received any study medication, and was based on the treatment allocated by the Interactive voice response system (IVRS) at randomization (as randomized). Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Gout flares
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 83
Gout flares | 1.23 (1.57) | 0.35 (0.67) | 0.34 (0.86)

2. Secondary Outcome: Number of Modified Gout Flares Per Participant From Day 1 to Day 113 (Week 16)
Description: Modified gout flare was defined using modified definition of a gout flare as participant-reported articular pain typical of a gout attack that was deemed to require treatment with anti-inflammatory therapy. Number of modified gout flares per participant were reported for this outcome measure.
Time Frame: Day 1 to Day 113 (Week 16)
Population: FAS that included all randomized participants who received any study medication, and was based on the treatment allocated by the IVRS at randomization (as randomized). Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Gout flares
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 83
Gout flares | 1.51 (1.87) | 0.62 (1.32) | 0.48 (0.99)

3. Secondary Outcome: Percentage of Participants With at Least One Flare From Day 1 to Day 113 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain; and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare was reported for this outcome measure.
Time Frame: Day 1 to Day 113 (Week 16)
Population: FAS that included all randomized participants who received any study medication, and was based on the treatment allocated by the IVRS at randomization (as randomized).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 84
percentage of participants | 56.1 | 25.6 | 20.5

4. Secondary Outcome: Percentage of Participants With at Least Two Flares From Day 1 to Day 113 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least two gout flares was reported for this outcome measure.
Time Frame: Day 1 to Day 113 (Week 16)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 84
percentage of participants | 32.9 | 8.5 | 6.0

5. Secondary Outcome: Number of Gout Flare Days Per Participant From Day 1 to Day 113 (Week 16)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flare days per participant was reported for this outcome measure.
Time Frame: Day 1 to Day 113 (Week 16)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 83
Gout flare days | 11.7 (21.0) | 4.30 (17.13) | 1.86 (5.80)

6. Secondary Outcome: Number of Gout Flare Days With Participant's Pain Score of 5 or More (From Daily Diary) Per Participant From Day 1 to Day 113 (Week 16)
Description: Participants were asked to complete a telephone diary by calling the IVRS daily beginning at the baseline visit (Day 1) through the follow-up visit (Day 141) and reported their general well-being, gout symptoms, and weekly study drug administrations. At the onset of pain from a gout flare, participants were to answer additional diary questions regarding their gout flare and had to continue daily flare assessments until they reported the flare had ended. If a flare occurred just prior to the follow-up visit (Day 141), participants were to continue completing the daily diary until the flare resolved. Gout flare pain was assessed on a scale from 0 to 10 (with 0=no pain and 10=severe pain) within the past 24 hours.
Time Frame: Day 1 to Day 113 (Week 16)
Population: FAS that included all randomized participants who received any study medication, and was based on the treatment allocated by IVRS at randomization (as randomized). Here, number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Number analyzed (Participants) | 82 | 82 | 83
Gout flare days | 4.28 (7.67) | 1.67 (8.43) | 0.88 (2.66)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational product
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the administration of first dose of study drug up to 35 days after the last dose of study drug).
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept ) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
Arm/Group | Placebo | Rilonacept 80 mg | Rilonacept 160 mg
Serious Adverse Events (participants affected / at risk) | 4/82 | 5/82 | 3/84
Other Adverse Events (participants affected / at risk) | 12/82 | 20/82 | 20/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Rilonacept 80 mg (N=82) | Rilonacept 160 mg (N=84)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Rilonacept 80 mg (N=82) | Rilonacept 160 mg (N=84)
Injection site erythema (General disorders) | 0 (0) | 6 (21) | 7 (20)
Influenza (Infections and infestations) | 6 (6) | 5 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (6) | 6 (6)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (3) | 6 (6) | 4 (5)
Headache (Nervous system disorders) | 2 (2) | 5 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.